CLINICAL TRIAL: NCT04498793
Title: Study of Tislelizumab Plus Chemotherapy vs Chemotherapy Alone as Perioperative Treatment in Participants With HER2 Negative Breast Cancer
Brief Title: Study of Tislelizumab Plus Chemotherapy vs Chemotherapy as Perioperative Treatment in Participants With HER2 Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Beijing Huanxing Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2474
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: HER2-negative Breast Cancer
MeSH Terms: interventions — tislelizumab; Taxes; Doxorubicin; Epirubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 group (Experimental): Participants receive tislelizumab every 3 weeks (Q3W) + nab-paclitaxel weekly x 4 cycles, followed by tislelizumab Q3W + (doxorubicin OR epirubicin) + cyclophosphamide Q3W x 4 cycles as neoadjuvant therapy prior to surgery; followed by 14 cycles of tislelizumab Q3W plus capecitabine (TNBC subtype) or endocrine therapy (Luminal subtype) as adjuvant therapy post-surgery.
  Each cycle is 21 days.
  Interventions: Biological: Tislelizumab; Drug: Nab paclitaxel; Drug: Doxorubicin; Drug: Epirubicin; Device: Cyclophosphamide
- Control group (Active Comparator): Participants receive nab-paclitaxel weekly x 4 cycles followed by (doxorubicin OR epirubicin) + cyclophosphamide Q3W x 4 cycles as neoadjuvant therapy prior to surgery; followed by capecitabine (TNBC subtype) or endocrine therapy (Luminal subtype) as adjuvant therapy post-surgery.
  Each cycle is 21 days.
  Interventions: Drug: Nab paclitaxel; Drug: Doxorubicin; Drug: Epirubicin; Device: Cyclophosphamide

INTERVENTIONS:
Biological: Tislelizumab — On Day 1 of the last seven cycles in the neoadjuvant and each cycle in the adjuvant phases of the study for a total of 21 cycles; intravenous (IV) infusion.
  Arms: PD-1 group
Drug: Nab paclitaxel — On Days 1 and 8 of Cycles 1-4 in the neoadjuvant phase of the study; IV infusion.
Drug: Doxorubicin — On Day 1 of Cycles 5-8 of the neoadjuvant phase of the study; IV injection.
Drug: Epirubicin — On Day 1 of Cycles 5-8 of the neoadjuvant phase of the study; IV injection.
Device: Cyclophosphamide — On Day 1 of Cycles 5-8 of the neoadjuvant phase of the study; IV infusion.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tislelizumab plus chemotherapy vs chemotherapy alone as perioperative treatment in participants who have triple negative HER2 negative breast cancer.

After a screening phase of approximately 28 days, each participant will receive neoadjuvant study treatment (Tislelizumab + Chemotherapy OR Chemotherapy) based on the randomization schedule for approximately 24 weeks (8 cycles). Each participant will then undergo definitive surgery 3-6 weeks after conclusion of the last cycle of the neoadjuvant study treatment.

After definitive surgery, each participant will receive adjuvant study treatment (routine adjuvant treatment +/- Tislelizumab) for approximately 42 weeks (14 cycles).

Following adjuvant study treatment, each participant will be monitored for safety, survival and disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of invasive breast cancer, cT1-T3, cN0-N3, cM0, HR+ (ER+ and/or PR+) HER2 negative or HR- (ER- and PR-) HER2 negative/triple negative breast cancer.
* Provides a core needle biopsy consisting of at least 2 separate tumor cores from the primary tumor at screening to the central laboratory.
* Immune active subtype revealed by multiplexed
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 performed within 10 days of treatment initiation.
* Demonstrates adequate organ function.

Exclusion Criteria:

* Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Has received prior chemotherapy, targeted therapy, or radiation therapy for breast cancer.
* Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death - ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g. CTLA-4, OX-40, CD137)
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (i.e. dosing exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or Hepatitis C.
* Has a known history of active tuberculosis.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has significant cardiovascular disease, such as: history of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last 6 months OR congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV or history of CHF NYHA Class III or IV.
* Pregnant or lactating women are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | Up to 30 weeks
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current American Joint Committee on Cancer (AJCC) staging criteria assessed by the local pathologist at the time of definitive surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Huanxing Cancer Hospital, Beijing, Beijing Municipality